CLINICAL TRIAL: NCT03005457
Title: A Low-cost Virtual Reality Gaming Platform for Neurorehabilitation of Hemiparesis
Brief Title: Pilot Study to Assess the Feasibility and Initial Efficacy of Therapist-as-consultant, Game-based CI Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Nationwide Children (Unknown)
Responsible Party: Principal Investigator, Lynne Gauthier , PhD, Assistant Prof. PM&R, Ohio State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 60047824
Record Dates: First submitted 2016-12-21; First posted 2016-12-29 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Stroke; Hemiparesis; Upper Extremity Dysfunction
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stroke (Experimental)
  Interventions: Behavioral: Hemiparesis Therapy with VR
- Hemiparesis other (Experimental)
  Interventions: Behavioral: Hemiparesis Therapy with VR

INTERVENTIONS:
Behavioral: Hemiparesis Therapy with VR — An in-home therapist-as-consultant model of CI therapy in which motor practice with shaping and the Motor Activity Log with problem solving were delivered via a custom avatar-based video game called Recovery Rapids

SUMMARY:
Pilot study to assess the feasibility and initial efficacy of therapist-as-consultant, game-based CI therapy. Pre/post study design. Participant received a target of 30 hours game-based motor intervention, 100 hours constraint of the less affected upper extremity, and 5 hours therapist consultation (including completion of a behavioral contract at the first study visit). Duration of intervention was 10 consecutive weekdays, with pre-treatment and post-treatment testing performed within 1 week prior to and 1 week post-intervention by an independent tester.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* Willing to comply with all study procedures and be available for the duration of the study
* Male or female aged > 17
* Preserved ability to comprehend English and participate in basic elements of the therapy
* Community-dwelling
* Experienced mild to moderate hemiparesis at least six months prior
* Can independently operate the gaming system (those with severe cognitive impairments can usually achieve this)
* Corrected vision of at least 20/70 as assessed by their ability to identify game objects on the monitor from 5 feet away

Exclusion Criteria:

* concurrent participation in other experimental upper extremity trials
* concurrent participation in other outpatient rehabilitation for their upper extremity
* Botox within the last 3 months (confound)
* near-normal motor function (9-hole Peg Test score above the 10th percentile of a normative sample)
* minimal nonuse (Motor Activity Log at baseline >2.5, Accelerometry > 60%)
* major medical issues that would interfere with study treatments or make intensive rehabilitation difficult to tolerate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in Motor Activity Log | Week 0 and Week 3
  Self-report measure of arm use for daily activities
Change in Wolf Motor Function Test | Week 0 and Week 3
  Objective measure of motor function in a laboratory setting

SECONDARY OUTCOMES:
Kinematic Data | Week 0 and Week 3
  Kinematic data recorded during game play
Brief Kinesthesia test | Week 0 and Week 3
  Clinical Assessment of sensation
Patient Health Questionnaire | Week 0 and Week 3
  Measures Depression
Strok Specific Quality of Life Scale | Week 0 and Week 3
  Quality of life measurement
Weschler Adult Intelligence Scale Symbol Seach | Week 0 and Week 3
  Cognitive processing speed assessment
Montreal Cognitive Assessment | Week 0 and Week 3
  Baseline cognitive screen
Survey | Week 0 and Week 3
  Survey on satisfaction with the intervention
Mitt Compliance | Week 0 and Week 3
  Hours of use
Total game-play time | Week 0 and Week 3
Gestures | Week 0 and Week 3
  Number of gestures of each type registered in game
Bilateral activity monitors | Week 0 and Week 3
  Objective measure of arm use
Action Research Arm Test (ARAT) | Week 0 and Week 3
  Asses Changes in Limb Function

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, 2154 Dodd Hall, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Will be shared upon publication acceptance.

REFERENCES:
- [Derived] Kelly KM, Borstad AL, Kline D, Gauthier LV. Improved quality of life following constraint-induced movement therapy is associated with gains in arm use, but not motor improvement. Top Stroke Rehabil. 2018 Oct;25(7):467-474. doi: 10.1080/10749357.2018.1481605. Epub 2018 Sep 22. PMID 30246613